CLINICAL TRIAL: NCT07140575
Title: Seamless Integration of Repetitive Transcranial Magnetic Stimulation (rTMS) for Youth Inpatients With Depression: A Feasibility Study
Brief Title: rTMS for Youth Inpatients With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Enoch Ng, Staff Psychiatrist and Associate Scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6604
Record Dates: First submitted 2025-07-31; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Major Depression Moderate; Feasibility Studies
Keywords: feasibility study; major depressive disorder; adolescent; youth; repetitive transcranial magnetic stimulation; neuromodulation; rTMS; accelerated; inpatient
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- repetitive transcranial magnetic stimulation (rTMS) (Experimental): twice daily rTMS (intermittent theta burst stimulation targeting the left dorsolateral prefrontal cortex)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — twice daily rTMS, intermittent theta burst stimulation targeting the left dorsolateral prefrontal cortex with a figure-8 coil

SUMMARY:
Youth aged 15-24 are likelier to have depression than all age groups in Canada. One-third of depressed youth do not respond to psychotherapy and/or antidepressant medications. A treatment called repetitive transcranial magnetic stimulation or rTMS has proven helpful in adolescents and young adults whose depressive symptoms have been difficult to treat with psychotherapy and/or antidepressants. Unfortunately, youth find rTMS difficult to access because it is not funded by the Ontario Health Insurance Plan, is typically only offered to adults, and the treatment schedule usually involves once-daily sessions, 5 days/week, for 4-6 weeks, which is associated with travel and opportunity costs e.g. missing school. This project looks at the feasibility of a new treatment pathway that allows youth with difficult-to-treat depression in hospital to receive rTMS twice-daily while engaging in on-unit schooling and therapeutic support. This "accelerated" way of providing rTMS is safe, has equal effectiveness to once-daily rTMS, and can shorten the time needed for treatment. This pathway is for youth already staying in hospital for difficult-to-treat depression or youth outside hospital who have difficult-to-treat depression that interferes with daily function to such a degree that they would benefit from staying in hospital. The investigators anticipate integrating rTMS and inpatient care for youth will be feasible, that it will be acceptable and accessible to youth and families, and there will be sufficient demand for this new treatment pathway. If successful, this project will inform care for youth with difficult-to-treat depression in Ontario and beyond.

ELIGIBILITY:
Inclusion Criteria:

* age 14-19 years
* primary diagnosis of major depressive disorder or of bipolar I or II disorder, current episode depressed with no psychotic or mixed features
* current episode of depression lasting at least 4 weeks
* failed ≥1 evidence-based psychotherapy or antidepressant
* have a GRID-HAMD-17 (17-item Hamilton Depression Rating Scale) score of ≥16 (moderate-severe range)
* currently an inpatient or suitable for an elective inpatient admission

Exclusion Criteria:

* lifetime diagnosis of a psychotic disorder, anorexia nervosa, bulimia nervosa diagnosis of a substance use disorder (except caffeine and tobacco) within the past year
* obsessive compulsive disorder or personality disorder that is the main source and driver of distress
* active psychosis and/or mania
* history of epilepsy or any other neurologic condition that includes a history of seizures
* use of medications that lower the seizure threshold
* pregnancy or nursing
* history of severe headaches within the previous year
* improvement in depressive symptom severity between screening and baseline by 25% or more
* inability to adhere to the protocol

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasible: 90% of the time, rTMS treatment will be started within 3 business days of a patient consenting during an existing inpatient stay or within 3 business days of the start of an elective inpatient stay | From enrollment to start of rTMS treatment, assessed for 8 weeks
  The investigators anticipate the treatment path will be feasible, operationalized as the ability to meet the following metric:
  Starting inpatient rTMS treatment within 3 business days of consenting during an existing inpatient stay or within 3 business days of the start of an elective inpatient stay - this metric will be met 90% of the time
Feasible: 90% completion of weekly Hamilton Depression Rating Scale during treatment by clinician | From start of rTMS treatment to end of rTMS treatment, assessed for 4 weeks
  The investigators anticipate the treatment path will be feasible, operationalized as the ability to meet the following metric:
  Completion of the clinician-administered 17-item Hamilton Depression Rating Scale weekly during rTMS treatment with 90% completion rate. The 17-item Hamilton Depression Rating Scale has a minimum score of 0 and maximum score of 52 with higher scores reflecting greater symptom burden.
Acceptable: 25% or lower drop-out rate from completing treatment | From enrollment to end of rTMS treatment, assessed for 12 weeks
  The investigators anticipate the treatment pathway will be acceptable to patients and families. Acceptability is operationalized as a 25% or lower drop-out rate from completing treatment.
Accessible: 90% of the time, suitability assessments for this treatment pathway will be completed within 2 business days for exiting inpatients and within 2 weeks for outpatients | From referral to suitability assessment and enrollment, assessed for 2 weeks
  The investigators the treatment pathway will be accessible to patients and families. Accessibility is operationalized as timelines of assessment: assessing referrals within 2 business days for existing inpatients and within 2 weeks (10 business days) for current outpatients. This metric will be met 90% of the time.
Demand: at least 30 youth will consent to being participants in this study | From referral to suitability assessment and enrollment, assessed for 2 weeks
  The investigators anticipate sufficient demand for this treatment pathway, operationalized as 30 youth consenting to being participants in this study. Alternatively, at least 30% of approached inpatient youth will consent to being participants in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No